CLINICAL TRIAL: NCT05566548
Title: The Importance of Bilirubin Molecular Species in Patients With Liver Cirrhosis Who Develop Hepatic Encephalopathy and Patients With Acute-on-chronic Liver Failure
Brief Title: Role of Bilirubin Molecular Species in Hepatic Encephalopathy and Acute-on-chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medica Sur Clinic & Foundation (Other)
Responsible Party: Principal Investigator, Nahum Méndez-Sánchez, Principal investigator, Medica Sur Clinic & Foundation
Other Study IDs: 2021-EXT-637
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure
Keywords: Bilirubin; Unconjugated bilirubin; Conjugated bilirubin; Bilirubin diglucuronide; Bilirubin monoglucuronide; ACLF; Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group of patients with liver cirrhosis and ACLF: This group will include patients with diagnosed liver cirrhosis regardless of the cause hospitalized and/or presenting to the emergency department for possible ACLF.
  With any etiology of liver cirrhosis including alcoholic liver disease (ALD), chronic hepatitis C virus (HCV), metabolism associated fatty liver disease (MAFLD) and autoimmune liver diseases.
  Interventions: Diagnostic Test: Liquid Chromatography-Mass Spectrometry Method to identify bilirubin molecular species
- Group of patients with liver cirrhosis compensated: This group will include patients with diagnosed liver cirrhosis, any etiology of liver cirrhosis including alcoholic liver disease (ALD), chronic hepatitis C virus (HCV), metabolism associated fatty liver disease (MAFLD) and autoimmune liver diseases.
  No previous episodes of ACLF and at the time of admission.
  Interventions: Diagnostic Test: Liquid Chromatography-Mass Spectrometry Method to identify bilirubin molecular species
- Group of healthy people: People who do not have any acute or chronic degenerative disease. Participation on a voluntary basis.
  Interventions: Diagnostic Test: Liquid Chromatography-Mass Spectrometry Method to identify bilirubin molecular species
- Group of patients with liver cirrhosis and hepatic encephalopathy: This group will include patients with diagnosed liver cirrhosis who develop hepatic encephalopathy graded according to West Haven.
  Interventions: Diagnostic Test: Liquid Chromatography-Mass Spectrometry Method to identify bilirubin molecular species

INTERVENTIONS:
Diagnostic Test: Liquid Chromatography-Mass Spectrometry Method to identify bilirubin molecular species — It will determine the concentration of the different molecular species of bilirubin and examine the pattern of increase present in patients with liver cirrhosis who develop hepatic encephalopathy and acute-on-chronic liver failure (ACLF) compared to other groups like patients with liver cirrhosis and healthy people.

SUMMARY:
It has been identified that impaired liver function, as occurs in patients with liver cirrhosis, prevents proper conjugation of glucuronic acid with bilirubin; as a result, unconjugated bilirubin accumulates in the blood, and conjugated bilirubin is markedly altered to form diglucuronides or monoglucuronides. However, in the development and progress of acute-on-chronic liver failure (ACLF) there is not enough information about these processes and the possible concentration levels that they can take.

Also Hepatic encephalopathy (HE) is a reversible complication, but with a high mortality rate in patients with acute or chronic liver failure, as well as a consequence of the formation of portosystemic shunts.

DETAILED DESCRIPTION:
Liver cirrhosis is a pathological diagnosis characterized by diffuse fibrosis, severe alteration of intrahepatic arterial and venous flow, portal hypertension, and, ultimately, liver failure. The prevalence of liver cirrhosis in the Mexican population depends on various factors, including gender, ethnic groups, and geographic regions, in addition to the nature, frequency, and time of acquisition of the main risk factors for cirrhosis, such as the hepatitis B virus, hepatitis C virus (HCV) in addition to non-alcoholic steatohepatitis, non-alcoholic fatty liver or alcoholic liver disease. Liver cirrhosis has been classified as decompensated or compensated. Decompensated liver cirrhosis occurs when there is gradual progression over months causing liver and extrahepatic organ failure. On the other hand, if it appears suddenly, in a short-term deterioration for days or several weeks after the defined triggering disease, it is known as Acute-on-chronic liver failure (ACLF). ACLF is a syndrome characterized by acute and severe liver abnormalities as a result of different types of lesions present in patients with underlying chronic liver disease or cirrhosis, but unlike decompensated cirrhosis, it has a high short-term mortality.

It is important to determine the prognosis of patients with ACLF, in a short period of time, in order to act appropriately and reduce the use of temporary liver support or liver transplantation, an important variable that is included in various scores that assess liver function in different scenarios such as the Child-Pugh score and Model for End-stage Liver Disease (MELD) systems.

Among liver cirrhosis complications, there is the Hepatic encephalopathy (HE) involves a wide range of neurocognitive and psychiatric abnormalities that can range from subclinical neurological deficits and disturbances in attention to coma. Diagnosis of hepatic encephalopathy can be made using the West Haven (WH) criteria, which are clinical criteria that evaluate the degree of neurological deterioration and divide hepatic encephalopathy into 5 grades (from grade 0 to grade 4), with grades 3 and 4 having a worse prognosis. In addition to these criteria, it can be diagnose based on psychometric tests such as the Portosystemic- Encephalopathy- Syndrome test (PSE) and psychophysiological tests, such as the Critical flicker frequency (CFF). Despite the existence of this evidence and the WH criteria, there is no quantitative parameter that can be used to diagnose the hepatic encephalopathy. In addition, although the quantification of ammonia levels is carried out in multiple centers as part of the protocol for diagnosing HE, there are numerous studies showing that ammonia levels cannot be used to diagnose or rule out the presence of HE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute-on-chronic liver failure (ACLF)
* Patients hepatic encephalopathy (HE)
* Any etiology of liver cirrhosis alcoholic liver disease (ALD), HCV, liver disease fatty liver associated with metabolism dysfunction (MAFLD) and diseases autoimmune liver
* With or without the existence of any precipitating event or medical complication: infection acute bacterial, consumption hepatitis severe alcoholic, variceal bleeding, drug-induced encephalopathy, ascites, coagulopathy, sepsis
* Any ACLF grade
* Any HE grade

Exclusion Criteria:

* Immunodeficiency virus infection human (HIV)
* Cholestatic liver disease,
* Past or current extrahepatic malignant tumor,
* Liver transplant,
* Other serious concomitant diseases heart, lung, kidney, or other organs
* Patients with metastatic hepatocellular carcinoma (HCC)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted in emergency room or hospitalized for liver cirrhosis with development of ACLF and hepatic encephalopathy. Also patients with liver cirrhosis compensated and healthy people.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Identify levels of Conjugated Bilirubin as Bilirubin monoglucuronide (BMG), bilirubin diglucuronide (BDG) and unconjugated bilirubin (UCB) in patients with acute-on-chronic liver failure | The serum sample will be taken at the moment of the first patient physician contact (admission, medical visit). The bilirubin measure will be done 24 hours after
  Identification and measured concentration of bilirubin molecular species through liquid chromatography-mass spectrometry (LC-MS)

SECONDARY OUTCOMES:
Comparison of the bilirubin levels of the different groups | It will be analyzed when all the results from the LC-MS are done. Approximately 5 months.
  The results of the groups will be compared among them to evaluate whether or not there is a change in the concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Nahum Mendez-Sanchez, MD, PhD, Study Director — Medica Sur Clinic & Foundation
Locations (1):
- Medica Sur Clinic & Foundation Organization, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karimzadeh P, Fallahi M, Kazemian M, Taslimi Taleghani N, Nouripour S, Radfar M. Bilirubin Induced Encephalopathy. Iran J Child Neurol. 2020 Winter;14(1):7-19. PMID 32021624
- [Background] Tapper EB, Rahimi RS. Low-Value Levels: Ammonia Testing Does Not Improve the Outcomes of Overt Hepatic Encephalopathy. Am J Gastroenterol. 2020 May;115(5):685-686. doi: 10.14309/ajg.0000000000000454. PMID 31714365
- [Result] Lopez-Velazquez JA, Chavez-Tapia NC, Ponciano-Rodriguez G, Sanchez-Valle V, Caldwell SH, Uribe M, Mendez-Sanchez N. Bilirubin alone as a biomarker for short-term mortality in acute-on-chronic liver failure: an important prognostic indicator. Ann Hepatol. 2013 Jan-2014 Feb;13(1):98-104. PMID 24378272
- [Result] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Result] Lee HA, Jung JY, Lee YS, Jung YK, Kim JH, An H, Yim HJ, Jeen YT, Yeon JE, Byun KS, Um SH, Seo YS. Direct Bilirubin Is More Valuable than Total Bilirubin for Predicting Prognosis in Patients with Liver Cirrhosis. Gut Liver. 2021 Jul 15;15(4):599-605. doi: 10.5009/gnl20171. PMID 33293481
- [Result] Tang L, Zhang M, Li X, Zhang L. Glucuronidated bilirubin: Significantly increased in hepatic encephalopathy. Prog Mol Biol Transl Sci. 2019;162:363-376. doi: 10.1016/bs.pmbts.2018.12.009. Epub 2019 Mar 6. PMID 30905463
- [Result] Bajaj JS, O'Leary JG, Tandon P, Wong F, Garcia-Tsao G, Kamath PS, Maliakkal B, Biggins SW, Thuluvath PJ, Fallon MB, Subramanian RM, Vargas HE, Lai J, Thacker LR, Reddy KR. Hepatic Encephalopathy Is Associated With Mortality in Patients With Cirrhosis Independent of Other Extrahepatic Organ Failures. Clin Gastroenterol Hepatol. 2017 Apr;15(4):565-574.e4. doi: 10.1016/j.cgh.2016.09.157. Epub 2016 Oct 5. PMID 27720916